CLINICAL TRIAL: NCT02624193
Title: Improving Treatment Adherence in HIV-Positive Youth Through Mindfulness Training
Brief Title: Health Improvement for Baltimore Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00093335; 1R01AT007888 (NIH)
Record Dates: First submitted 2015-06-10; First posted 2015-12-08 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: HIV; Adolescent Development; Adolescent Behavior; Medication Adherence
Keywords: Treatment Adherence; Mental Health; Well-being; Emerging Adults; Youth
MeSH Terms: conditions — Adolescent Behavior; Medication Adherence; Treatment Adherence and Compliance; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBSR Program (Experimental): MBSR Program:
  The MBSR intervention is a nine-week program designed to cultivate mindfulness, a focused non-judgmental awareness of the present moment. It consists of eight 2-hour weekly sessions and one 3-hour retreat and the content includes three main components: 1) material related to mindfulness, meditation, yoga, and the mind-body connection; 2) experiential practice of mindful meditation (sitting, lying down, walking), gentle mindful yoga, and "body scan" during group meetings and encouragement of home practice; and 3) group discussion focused on problem-solving related to barriers to effective practice. HIV disease will not be discussed as a group topic, unless it is brought up by participants.
  Interventions: Behavioral: MBSR Program
- HT Program (Placebo Comparator): Healthy Topics Program:
  The health education program "Healthy Topics" (HT) will serve as an attention control group. The HT program is focused on providing age-appropriate health information and education. There is minimal content overlap in the MBSR and HT programs regarding self-care and healthy eating; however, the style, structure, and content of the MBSR and HT programs are distinct. HT participants will receive no training in MBSR or meditation. Topics covered include physical activity, nutrition, managing weight, building health, personal care, understanding adolescence, tobacco, alcohol, and other drugs. HIV disease will not be discussed as a group topic, unless it is brought up by participants.
  Interventions: Behavioral: HT Program

INTERVENTIONS:
Behavioral: MBSR Program — Mindfulness-based stress reduction, as described previously.
  Other Names: Mindfulness Program
  Arms: MBSR Program
Behavioral: HT Program — Health education curriculum, as described previously
  Other Names: Healthy Topics Program
  Arms: HT Program

SUMMARY:
Preliminary data from the investigators' National Center for Complementary and Alternative Medicine (NCCAM)-funded R21 on mindfulness-based stress reduction (MBSR) in HIV-infected youth suggest an association between mindfulness and improved self-regulation and medication adherence. This randomized, controlled trial will help the investigators to better understand the specific impact of MBSR on HIV medication and treatment adherence in HIV-infected youth, and the efficacy of MBSR in the amelioration of stress and improved self-regulation.

DETAILED DESCRIPTION:
Despite remarkable advances in HIV medication effectiveness, adherence to HIV treatment recommendations is alarmingly poor, resulting in preventable morbidity and mortality. It is estimated that 26-72% of HIV-infected adolescents are non-adherent to their HIV medications and 22-33% are non-adherent with scheduled health care visits. HIV treatment non-adherence puts individuals at markedly increased risk for illness related to HIV itself and a variety of opportunistic infections, as well as at increased risk of spreading HIV.

Preliminary data from the investigators' NCCAM-funded R21 on mindfulness-based stress reduction (MBSR) in HIV-infected youth suggest an association between mindfulness and improved medication adherence, as well as enhanced self-regulatory processes (coping, psychological function, and cognitive function). This two-armed randomized, controlled trial will help the investigators to better understand the specific impact of MBSR on HIV medication and treatment adherence in HIV-infected youth, and the efficacy of MBSR in the amelioration of stress and improved self-regulation.

The aims of the study are as follows:

Primary Objective

Investigators hypothesize that MBSR vs. active control program (HT) participation will be associated with:

• (H1) Improved HIV medication adherence (self-report validated by HIV viral load) at 3 months, 6 months, and 12 months

Secondary Objectives

Investigators also hypothesize that MBSR vs. active control program (HT) participation will be associated with:

* (H2) Improved coping at 3, 6, and 12 months
* (H3) Improved psychological functioning at 3, 6, and 12 months
* (H4) Improved cognitive functioning at 3, 6, and 12 months

Investigators will also explore:

* associations (and potential mediation) among mindfulness, self-regulation, and HIV medication adherence and
* using qualitative methods, experience with MBSR, HIV treatment adherence, as well as reasons for non-participation in the study and non-attendance of program sessions to inform future implementation planning.
* gender differences in the effects of MBSR versus HT on emotion regulation and physiological responses to stressful stimuli.

ELIGIBILITY:
Inclusion Criteria:

* 13-24 years of age
* English speaking
* Receiving care at the adolescent outpatient clinics at Johns Hopkins Children's Center (JHCC/University of Maryland Medical Center (UMMC)/Moore Clinic
* Positive for HIV and aware of his/ her status
* Prescribed anti-retroviral therapy (ART)
* Able to attend and participate in the 9 week program sessions

Exclusion Criteria:

* patient currently exhibits significant psychological, developmental, or behavioral issues as assessed by the site clinical staff
* participated in a previous MBSR program or studies

Exclusion Criteria for supplement study:

• patient is transgender

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2013-04; Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Treatment Adherence | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on treatment adherence as measured by the Adolescent Medicine Trials Network (ATN) HIV Medication Adherence self-report measure, as well as CD4 and viral load counts pulled from the participant's medical record. The measure and medical record data collection takes place at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.

SECONDARY OUTCOMES:
NIH Emotion Measures Questionnaire | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on emotion regulation measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up. Specific NIH emotion measures are: meaning & purpose, positive affect, anger, fear, perceived hostility, sadness.
Illness Cognition (IC) Scale | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on thoughts of illness measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Difficulties in Emotion Regulation Scale (DERS) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on issues in emotion regulation measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Mindful Acceptance and Awareness Scale (MAAS) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on mindfulness measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Five Facet Mindfulness Questionnaire (FFMQ) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on multiple aspects of mindfulness measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Differential Emotions Scale (DES) - selected items | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on frequency of emotions (specifically, self-hostility, shame, shyness, and guilt) measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
State-Trait Anger Expressivity Inventory (STAXI) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on anger expression measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Children's PTSD Symptom Severity Checklist (CPSS) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on trauma symptoms measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Compassion Scale | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on self-compassion measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Perceived Stress Scale (PSS) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on perceived stress measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Sex Risk Scale | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on risky sexual behavior measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Lesbian & Gay Identity Scale (LGIS) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on self-acceptance of lesbian/gay/bisexual identity measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
General Health Assessment | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on general health measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Youth Quality of Life scale (YQOL) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on quality of life measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Brief COPE Questionnaire | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on coping measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Children's Response Style Questionnaire (CRSQ) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on coping responses measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Das-Naglieri Cognitive Assessment System (CAS) | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on cognitive functioning measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.
Emotion Stroop Task | Baseline, and follow up at 3, 6, and 12 months
  Assessment of impact of MBSR versus HT on emotion-based cognitive functioning measured at baseline, post-program (3-month follow-up), 6-month follow-up, and 12-month follow-up.

OTHER OUTCOMES:
Berkeley Expressivity Questionnaire (BEQ) | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on emotion expressivity (by gender) measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
Children's Emotion Management Scales (CEMS) | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on management of anger, sadness, happiness, pride, and worry (by gender) measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
Differential Emotions Scale (DES) | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on the frequency of emotions, specifically disgust, joy, sadness, surprise, contempt, interest, fear, and anger, (by gender) measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
Emotion Regulation Questionnaire (ERQ) | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on emotion regulation (by gender) measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
Emotion Approach Coping Scale (EAC) | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on emotion approach coping (by gender) measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
Flanker Inhibitory Control and Attention Test Age 12+ v2.0 | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on stress response, and inhibitory control and attention (by gender) measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
List Sorting Working Memory Test Age 7+ v2.0 | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on stress response, and working memory (by gender) measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
Dimensional Change Card Sort Test Age 12+ v2.0 | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on stress response, and cognitive flexibility, measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
Picture Sequence Memory Test Age 8+ (Form A) v2.0 | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on stress response, and episodic memory measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.
Heart Rate Variability (HRV) | Baseline, and follow up at 3, 6, and 12 months
  For those selected to be in the supplement study, assessment of impact of MBSR versus HT on stress response measured at baseline, post-program (3-month follow up), 6-month follow-up, and 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Sibinga, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Harriet Lane Clinic, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No